CLINICAL TRIAL: NCT01348464
Title: Transumbilical Single Port Laparoscopic Appendectomy Versus Conventional Laparoscopic Appendectomy in Adult Patients: A Prospective Randomized Control Study
Brief Title: A Trial on Laparoscopic Appendectomy Versus Single Port Appendectomy
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Won-Suk Lee, Assistant prof, Gachon University Gil Medical Center
Other Study IDs: girba2339
Record Dates: First submitted 2011-04-29; First posted 2011-05-05 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Acute Appendicitis
Keywords: appendectomy; appendicitis; laparoscopic surgery
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lifestyle, wound satisfaction: single site access three site access for appendectomy
  Interventions: Procedure: single port appendectomy, three port appendectomy

INTERVENTIONS:
Procedure: single port appendectomy, three port appendectomy — visual analog scale. questionnaire on wound satisfaction
  Other Names: Pain scale; Satisfactory score; complication rate

SUMMARY:
The aim of this study is to compare patients who undergone single-port access laparoscopic appendectomy to those who underwent conventional three-port laparoscopic appendectomy (TPLA) in a prospective randomized trial

DETAILED DESCRIPTION:
* primary objective

  1. complication rate
* secondary objectives

  1. satisfaction rate
  2. pain scale difference

ELIGIBILITY:
Inclusion Criteria:

* age 5~85 years
* any patient diagnosed with acute appendicitis on appendix sonography or abdominopelvic CT
* Patient performance status(PS) with greater than 80 or more on Karnofsky PS
* Give written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

* Pregnant or lactating
* Serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease
* History of Previous cytotoxic chemotherapy, radiotherapy or immunotherapy, for the currently treated cancer
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohorts will be the residents of Incheon, Korea
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-03; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Complication rate | participants will be followed for the duration of hospital stay, an expected average of 24 weeks
  observe complication caused by both procedures

SECONDARY OUTCOMES:
patient satisfaction | participants will be followed for the duration of hospital stay, an expected average of 24 weeks
  Questionarire is given to the patients on postoperative 3days, 1month, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Won-Suk Lee, MD, Principal Investigator — Gachon Univ. Gil Medical Center
Locations (1):
- Gachon Univ., Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Background] Raakow R, Jacob DA. Initial experience in laparoscopic single-port appendectomy: a pilot study. Dig Surg. 2011;28(1):74-9. doi: 10.1159/000322921. Epub 2011 Feb 4. PMID 21293135
- See also: laparoscopic surgery teaching site — http://websurg.com/